CLINICAL TRIAL: NCT02332395
Title: The Evaluation of Postoperative Pain After Emergency and Elective Caesarean Section Operations
Brief Title: The Evaluation of Postoperative Pain After Caesarean Section
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assistant Professor, MD, Tokat Gaziosmanpasa University
Other Study IDs: 13-KAEK-226
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Pain
Keywords: pain; pain catastrophizing; cesarean section
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Emergency caesarean section: patients whose underwent emergency caesarean section operation
- Elective caesarean section: patients whose underwent elective caesarean section operation

SUMMARY:
The aim of this study is to determine the effect of surgical priority either emergency or elective on postoperative pain in caesarean section operations. Patients whose undergo caesarean section operation are included into this study. Patients will invite to complete the Pain Catastrophizing Scale questionnaire in preoperative period. The patients will be divided into two groups in terms of applied surgical priority whether emergency or elective. After caesarean section, patient controlled analgesia is used for pain relief. And the intensity of pain will be measured by using numerical rating scale.

DETAILED DESCRIPTION:
Pain is the main problem of postoperative period. Postoperative analgesic consumption can be associated with physical and psychological condition of the individual. This study is aimed to investigate the effect of surgical priority either emergency or elective on postoperative pain in caesarean section operations.

Patients are invited to complete the pain catastrophizing scale questionnaire in preoperative period.

A total of 100 patients will be included into the study. Patients are divided into two groups in terms of surgical priority whether emergency or elective. Spinal or general anesthesia will be performed to the patients. In postoperative period, patient controlled analgesia will be applied for pain relief and numerical rating scale is used to determine the pain intensity in 1st, 2nd, 6th, 12th, 24th hours. The analgesic consumption in 24 hours will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists score of 1 or 3 and 1-Emergency or 3-Emergency

Exclusion Criteria:

* Patients whose not to participate
* Patients whose have communication problems
* Patients whose have been using antipsychotic or antidepressant drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: individuals whose underwent caesarean section operation in terms of surgical priority whether emergency or elective
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Total amount of analgesics | 24 hours

SECONDARY OUTCOMES:
numerical rating scale | 24 hours
pain catastrophizing scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Ass.Prof, MD, Principal Investigator — Gaziosmanpasa University, Medical Faculty, Department of Anesthesiology and Reanimation
Locations (1):
- Gaziosmanpasa University, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Taşdemir A, Erakgün A, Nuri Deniz M, ÇertuğA . Preoperatif Bilgilendirme Yapılan Hastalarda Ameliyat öncesi ve Sonrası Anksiyete Düzeylerinin State-Trait Anxiety Inventory Test ile Karşılaştırılması. Turkish Journal Anaesthesiology and Reanimation 41(2): 44-9, 2013.
- [Background] Kırdemir P, Özorak Ö. Postoperatif Ağrı ve Analjezik İhtiyacı Preoperatif Dönemde Tahmin Edilebilir mi? Turkiye Klinikleri Journal of Medical Sciences 31(4):951-9, 2011.
- [Background] Hüseyinoğlu Ü, Ülker K, Temur İ, Kütük M. Elektif Sezaryen Doğum Sonrası Postoperatif Ağrı Gideriminde Meperidin ve Tramadolün Karșılaștırılması: Bir Prospektif Randomize Çalıșma. Kafkas Journal of Medical Sciences 1(2):53-56, 2011.